CLINICAL TRIAL: NCT06642415
Title: Effect Of High Magnification On Quality Of Life And Success After Endodontic Microsurgery: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jyoti Dnyaneshwar Nadekar
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Periapical Lesion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sham piezoelectric setup for patients undergoing conventional surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loupes group (Active Comparator): Surgery performed under loupes
  Interventions: Procedure: Surgery under loupes; Procedure: surgery performed under microscope
- Microscope group (Experimental): Surgery performed under microscope
  Interventions: Procedure: Surgery under loupes; Procedure: surgery performed under microscope

INTERVENTIONS:
Procedure: Surgery under loupes — surgery performed under loupes
Procedure: surgery performed under microscope — surgery performed under microscope

SUMMARY:
Effect of high magnification on quality of life and success after endodontic surgery: a randomized controlled trial"

DETAILED DESCRIPTION:
: Residual infection in untreated canal space is one of the most common cause of post treatment apical periodontitis. The prevalence of post treatment apical periodontitis has been reported to be 60% to 80%. Endodontic microsurgery and root resection removes the inaccessible apical ramifications and ensures adequate sealing of apical communication. Magnification has been recommended for better visualization of apical terminus. Various case reports and retrospective studies have reported higher success of apical surgery when magnification devices have been used as an adjunct to periapical surgery (setzer 2010, tsesis 2006, bud 2020). However, there are very few prospective studies and there is heterogeneity in data in terms of type of magnification used and there are very few studies comparing different magnification devices.

To the best of our knowledge no randomized controlled trial has been done on the periapical surgery of maxillary anterior teeth which compares the effect of magnification by microscope versus loupes, hence the aim of this study is to assess the quality of life and success after endodontic surgery using with or without magnification.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age of 18-55 with the diagnosis of persistent symptomatic apical periodontitis in previously treated teeth with radiographic evidence of periapical radiolucency (≥ 5 mm). (Bharathi et al 2021) Tooth with a peri radicular lesion of strictly endodontic origin and unrestorable by nonsurgical retreatment. ASA-1 patients according to the classification of the American Society of Anesthesiologists).

Exclusion Criteria:

Patients with systemic diseases (diabetes mellitus, uncontrolled hypertension grade III, hepatic/renal disease, or systemic bleeding disorders) Combined endodontic-periodontic lesions Pregnancy

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment | till 7 days after surgery
  To determine the quality of life after endodontic microsurgery with high and low magnification using modified version of sugars et al and OHIP by tsesis et al. assessed by 5-point Likert scale till 1 week.
Healing assessment | After 6 months and 12 months
  2D radiographic healing was assessed by the criteria followed by RUD et al and MOLVEN et al , 3D CBCT healing was assessed by modified PENN'S criteria

SECONDARY OUTCOMES:
Pain assessment | till 7 postoperative days
  Pain assessment by VAS (0 - 100), where 0 is no pain and 100 is worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India